CLINICAL TRIAL: NCT05618613
Title: An Open-Label, Phase 1b-2 Study of Elacestrant, in Combination With Onapristone in Patients With Estrogen Receptor-Positive, Progesterone Receptor-Positive, HER2-negative Advanced or Metastatic Breast Cancer (ELONA)
Brief Title: Study of Elacestrant in Combination With Onapristone in Patients With Advanced or Metastatic Breast Cancer
Acronym: ELONA
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to discontinue onapristone development.
Sponsor: Context Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONA-XR-103
Record Dates: First submitted 2022-11-03; First posted 2022-11-16 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — elacestrant; RAD1901; onapristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Elacestrant / Onapristone (Experimental): Elacestrant and Onapristone combination
  Interventions: Drug: Elacestrant; Drug: Onapristone

INTERVENTIONS:
Drug: Elacestrant — Elacestrant 200mg, 300mg, or 400mg once daily oral dosing in cycles of 28 days.
  Other Names: RAD1901
Drug: Onapristone — Onapristone 40mg or 50mg twice daily oral dosing in cycles of 28 days.

SUMMARY:
This is a multicenter, Phase 1b-2 study of elacestrant in combination with onapristone in patients with advanced/metastatic ER+/PgR+/HER2- breast cancer.

DETAILED DESCRIPTION:
This is a multicenter, phase 1b-2 trial. The phase 1b part of the trial is open label and aims to determine the recommended Phase 2 dose (RP2D) of onapristone and elacestrant when administered together. The Phase 2 part of the trial will evaluate the efficacy and safety of this combination in patients with ER+/PgR+/HER2- advanced/metastatic breast cancer after prior therapy with a CDK4/6 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. Women or men aged ≥18 years, at the time of informed consent signature. Note: Pre- and peri-menopausal women must receive goserelin for at least one month prior to initiating trial therapy, during the trial, and for at least one month after end of trial therapy. Men must receive triptorelin for at least one month prior to initiating trial therapy, during the trial and for at least one month after end of trial therapy.
2. Histopathologically or cytologically confirmed ER+, PgR+, HER2-, breast cancer, per local laboratory, as per the American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines (Allison et al, 2020). Note: In the context of this trial, ER and PgR status will be considered positive if ≥10% of tumor cells demonstrate positive nuclear staining by immunohistochemistry.
3. At least one measurable lesion as per RECIST version 1.1. Note: Patients with stable brain or subdural metastases are allowed if the patient has completed local therapy and has discontinued the use of corticosteroids for at least 4 weeks before starting treatment in this study. Any signs (e.g., radiologic) or symptoms of brain metastases must be stable for at least 4 weeks before starting study treatment.
4. Prior therapy with an aromatase inhibitor or fulvestrant + a CDK4/6 inhibitor in the metastatic setting or in the adjuvant setting if within 12 months of last dose of adjuvant therapy. Note: Prior therapy with everolimus is allowed.
5. ECOG performance status of 0 or 1.
6. Patient has adequate bone marrow and organ function, as defined by the following laboratory values:

   1. Absolute neutrophil count (ANC) ≥1.5 × 109/L,
   2. Platelets ≥100 × 109/L,
   3. Hemoglobin ≥9.0 g/dL,
   4. Potassium, sodium, calcium (corrected for serum albumin), and magnesium CTCAE grade ≤1,
   5. Cockcroft-Gault-based creatinine clearance ≥50 mL/min. Note: Creatinine clearance (male) = ([140-age in years] × weight in kg)/ ([serum creatinine in mg/dL] × 72) Creatinine clearance (female) = (0.85 × [140-age in years] × weight in kg)/ ([serum creatinine in mg/dL] × 72),
   6. Serum albumin ≥3.0 g/dL (≥30 g/L),
   7. In absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0 × ULN. If the patient has liver metastases, ALT and AST ≤5 × ULN,
   8. Total serum bilirubin <1.5 × ULN except for patients with Gilbert's syndrome who may be included if the total serum bilirubin is ≤3.0 × ULN or direct bilirubin ≤1.5 × ULN.

Exclusion Criteria:

1. Active or newly diagnosed CNS metastases, including meningeal carcinomatosis.
2. Breast cancer treatment-naïve patients in the metastatic setting.
3. Prior therapy with elacestrant, onapristone, or chemotherapy in the metastatic setting.
4. Patient has a concurrent malignancy or history of invasive malignancy within 3 years of enrollment, with the exception of basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix that has completed curative therapy.
5. Uncontrolled significant active infections.

   1. Patients with hepatitis B virus (HBV) and/or hepatitis C virus (HCV) infection must have undetectable viral load during screening.
   2. Patients known to be HIV+ are allowed as long as they have undetectable viral load at baseline.
6. Major surgery within 4 weeks before starting trial therapy.
7. Inability to take oral medication, or history of malabsorption syndrome or any other uncontrolled gastrointestinal condition.
8. Females of childbearing potential who:

   1. Within 28 days before study entry, did not use a highly effective method of contraception.
   2. Do not agree to use a highly effective method of contraception throughout the entire study period and for 28 days after trial therapy discontinuation.
9. Males who do not agree to abstain from donating sperm, or to use a highly effective method of contraception, during the course of the treatment period and for 28 days thereafter.
10. Known intolerance to either study drug or any of the excipients.
11. Patient is currently receiving or received any of the following medications prior to first dose of trial therapy:

    1. Known strong or moderate inducers or inhibitors of cytochrome P450 (CYP) 3A4 within 14 days or 5 half-lives, whichever is shorter, (Refer to http://medicine.iupui.edu/clinpharm/ddis/),
    2. Herbal preparations/medications within 7 days. These include, but are not limited to, St. John's wort, kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng.
    3. Investigational anti-cancer therapy with 21 days or 5 half-lives, whichever is shorter.
    4. Vaccination, including but not limited to vaccination against COVID-19, during the 7 days prior to randomization.
12. Evidence of ongoing alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Determine the recommended Phase 2 dose (RP2D) of the combination of onapristone and elacestrant (Phase 1). | 9 months
Evaluate the efficacy of elacestrant in combination with onapristone in terms of objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors [RECIST] version 1.1 (Phase 2). | 1.5 years
  Proportion of patients achieving a best overall response of confirmed partial or complete response (PR+CR).

SECONDARY OUTCOMES:
Characterize the AEs of elacestrant in combination with onapristone. | 21 months
  Characterize the AEs of elacestrant in combination with onapristone.
Characterize the serious adverse events (SAEs) of elacestrant in combination with onapristone. | 21 months
  Characterize the serious adverse events (SAEs) of elacestrant in combination with onapristone.
Characterize the safety in terms of changes in clinical laboratory values of elacestrant in combination with onapristone. | 21 months
  Characterize the safety in terms of changes in clinical laboratory values of elacestrant in combination with onapristone.
Characterize the safety in terms of changes in vital sign measurements of elacestrant in combination with onapristone. | 21 months
  Characterize the safety in terms of changes in vital sign measurements of elacestrant in combination with onapristone.
Characterize the safety in terms of changes in ECG parameters of elacestrant in combination with onapristone. | 21 months
  Characterize the safety in terms of changes in ECG parameters of elacestrant in combination with onapristone.
Evaluate the area under the plasma concentration-time curve over the dosing interval of elacestrant as well as onapristone and their metabolites (Phase 1). | 9 months
  Evaluate the area under the plasma concentration-time curve over the dosing interval of elacestrant as well as onapristone and their metabolites (Phase 1).
Evaluate the maximum plasma concentration (Cmax) of elacestrant as well as onapristone and their metabolites (Phase 1). | 9 months
  Evaluate the maximum plasma concentration (Cmax) of elacestrant as well as onapristone and their metabolites (Phase 1).
Evaluate the time of the maximum observed plasma concentration (Tmax) of elacestrant as well as onapristone and their metabolites (Phase 1). | 9 months
  Evaluate the time of the maximum observed plasma concentration (Tmax) of elacestrant as well as onapristone and their metabolites (Phase 1).
Evaluate the trough concentration of elacestrant as well as onapristone and their metabolites (Phase 1). | 9 months
  Evaluate the trough concentration of elacestrant as well as onapristone and their metabolites (Phase 1).
Evaluate duration of response. | 3 years
  Time from the date of the first documented CR/PR until first documentation of disease progression or death, whichever comes first.
Evaluate clinical benefit rate. | 3 years
  Proportion of subjects achieving a best overall or complete response, or durable stable disease (duration is at least 23 weeks).
Evaluate progression-free survival. | 3 years
  Time from the date of the first dose to the date of the first documentation of disease progression or death, whichever occurs first.
Evaluate overall survival. | 3 years
  Time from first dose date to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Cancer Treatment Centers of America - Western Regional Medical Center, Phoenix, Arizona
  - Cancer Treatment Centers of America - Midwestern Regional Center, Zion, Illinois
  - Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No